CLINICAL TRIAL: NCT04236583
Title: Improving the Hospital-to-Home Transition Through Post-Discharge Virtual Visits in Primary Care
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Per IRB COVID-19 guidance on conducting human subjects research
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-09020793
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Telehealth
Keywords: Video Visits; Virtual Visits; Telehealth
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth (Experimental): Eligible patients will be given the option to consent to having one virtual visit with their primary care physician within four weeks after discharge from the hospital. Usual follow-up care will occur during this visit.
  Interventions: Other: Telehealth

INTERVENTIONS:
Other: Telehealth — Post-discharge virtual visit
  Other Names: Video Visits

SUMMARY:
The purpose of this study is to test a new process for having a virtual visit with a primary care doctor after discharge from the hospital, instead of an in-person visit.

DETAILED DESCRIPTION:
The goal of this project is to fully develop the protocol for identifying patients who would benefit from a virtual visit and develop the protocol for implementing the virtual visit. The value of this project is that the results will provide ample preliminary data for a future randomized controlled trial to determine the effectiveness of the intervention. This project will have an intervention group only. The hypothesis is that the intervention can be implemented in a way that is feasible and acceptable to providers and patients.

ELIGIBILITY:
Inclusion Criteria:

* Medical inpatients, age >=18, with an existing WCIMA attending as his or her PCP
* Patients with disposition to home
* Medically appropriate for a video visit (as determined by inpatient attending)
* Patients or caregivers must be able to enroll in MyChart before discharge, must be capable of using the Weill Cornell Connect app to do a video visit at home using broadband access or the equivalent (must own a device compatible with the app, e.g.

smartphone or tablet)

* English speaking
* Cognitively able to participate or Caregiver must be able to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients meeting inclusion criteria over the study period out of all patients being discharged over the same time period | 6 months post-intervention
Proportion of patients who consent to participate out of all those found to be eligible | 6 months post-intervention
Proportion of patients who successfully schedule video visits out of all of those who consent | 6 months post-intervention
Proportion of patients who successfully complete video visit out of all of those who scheduled | 6 months post-intervention

SECONDARY OUTCOMES:
Patient satisfaction with the video visit | Within one month post-intervention
  Based on a previously validated instrument (Parmanto et. al, Int J Telerehab 2016 Spring; 8(1): 3-10). Measured through 5-point likert scale,free response, multiple choice, and yes/no questions.
Physician satisfaction with the video visit | Within one month post-intervention
  Measured through multiple choice, yes/no, and free-response (only asked if specific responses are received) questions.
Number of in-person visits instead of or in addition to video visit | 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sanjai Sinha, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No